CLINICAL TRIAL: NCT01561560
Title: Clinical Evaluation of Two Daily Disposable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-347-C-019
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
Keywords: DAILIES TOTAL1; contact lenses; myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAILIES TOTAL1, then TRUEYE (Other): Delefilcon A contact lenses worn first, followed by narafilcon A contact lenses. Each product was worn bilaterally on a daily wear, daily disposable basis for two weeks.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses
- TRUEYE, then DAILIES TOTAL1 (Other): Narafilcon A contact lenses worn first, followed by delefilcon A contact lenses. Each product was worn bilaterally on a daily wear, daily disposable basis for two weeks.
  Interventions: Device: Delefilcon A contact lenses; Device: Narafilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — CE-marked, silicone hydrogel, soft contact lenses for daily wear, daily disposable use, worn bilaterally for two weeks in either Period One or Period Two
  Other Names: DAILIES TOTAL1®
Device: Narafilcon A contact lenses — CE-marked, silicone hydrogel, soft contact lenses for daily wear, daily disposable use, worn bilaterally for two weeks in either Period One or Period Two
  Other Names: 1-DAY ACUVUE® TRUEYE™

SUMMARY:
The purpose of this crossover study was to evaluate the end-of-day comfort of two commercially available, daily disposable, silicone hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Sign written Informed Consent Document.
* Currently wearing soft contact lenses in both eyes and identified as symptomatic based on questionnaire responses.
* Currently wearing either daily disposable contact lenses or weekly/monthly replacement contact lenses.
* Able to achieve visual acuity of at least 6/7.5 in each eye with study lenses in the available parameters.
* Willing to wear study lenses for at least eight hours per day and at least five days per week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has not worn contact lenses before.
* Currently wearing DAILIES TOTAL1 or 1-DAY ACUVUE TRUEYE contact lenses.
* Any systemic or ocular disease or disorder that would negatively affect the conduct or outcome of the study.
* Ocular surgery/trauma within the last six months.
* Topical ocular or systemic use of antibiotics within seven days of enrollment.
* Pregnant or nursing women.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Girault, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two study centers in Finland, three study centers in German, and three study centers in the UK.
Pre-assignment Details: Of the 123 participants enrolled, two were excluded prior to randomization. This reporting group includes all participants enrolled and exposed to Test Article (121).
Period: First Two Weeks of Wear
Arm/Group | DAILIES TOTAL1, Then TRUEYE | TRUEYE, Then DAILIES TOTAL1
Started | 60 | 61
Completed | 60 | 59
Not Completed | 0 | 2
Not completed — Time/job conflict | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Two Weeks of Wear
Arm/Group | DAILIES TOTAL1, Then TRUEYE | TRUEYE, Then DAILIES TOTAL1
Started | 60 | 59
Completed | 60 | 58
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled and exposed to Test Article
Groups:
- OVERALL: Delefilcon A contact lenses and narafilcon A contact lenses worn in randomized order. Each product was worn bilaterally on a daily wear, daily disposable basis for two weeks.
Arm/Group | OVERALL
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: End-of-day Comfort
Description: End-of-day comfort was interpreted and reported by the participant on a questionnaire as a single, retrospective measurement of two weeks of wear. Participants were asked, "Please rate the study lenses you have been wearing the in the following area: End-of-day comfort" and recorded their response on a continuous 1-10 Likert scale (1=poor and 10=excellent).
Time Frame: Week 2
Population: This reporting group includes all participants who finished the study, minus any major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- DAILIES TOTAL1: Delefilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for two weeks
- TRUEYE: Narafilcon A contact lenses worn in both eyes on a daily wear, daily disposable basis for two weeks
Arm/Group | DAILIES TOTAL1 | TRUEYE
Number analyzed (Participants) | 116 | 116
Units on a scale | 8.3 (1.91) | 6.6 (2.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all participants enrolled and exposed to Test Article.
Description: An adverse event was defined as an event that caused, or had the potential to cause, unexpected or unwanted effects involving the safety of device users (including patients) or other persons.
Arm/Group | DAILIES TOTAL1 | TRUEYE
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/121
Other Adverse Events (participants affected / at risk) | 0/119 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data should not be disclosed to any third party for a period of three years after the termination of the study without prior written consent.